CLINICAL TRIAL: NCT06944860
Title: Microbial Adherence, Surface Roughness, Effectiveness and Impact on Patients Between Conventional and 3D Printed Twin Block Appliances: An Open-Label Prospective Clinical Trial
Brief Title: Microbial Adherence, Surface Roughness, Effectiveness and Impact on Patients Between Conventional and 3D Printed Twin Block Appliances
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Wan Nurazreena Wan Hassan, Associate Professor, Department of Paediatric Dentistry & Orthodontics, Faculty of Dentistry Universiti Malaya, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2106613/2; IIRG002-2022HWB (Other Grant/Funding Number: Impact-Oriented Interdisciplinary Research Grant Programme); UMG034E-2025 (Other Grant/Funding Number: Universiti Malaya Dental Postgraduate Research Fund)
Record Dates: First submitted 2025-04-06; First posted 2025-04-25 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Orthodontic Appliances, Removable; Orthodontic Appliance Complication; Class II Malocclusion, Division 1
Keywords: Twin block appliance; Microbial adherence; Surface roughness; Effectiveness; Oral Health Related Quality of Life (OHRQoL)
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Intervention Model Description: Baseline characteristics - newly constructed conventional Twin Block appliances and 3D printed Twin Block appliances will be tested for microbial analysis, surface roughness, effectiveness and the impact on the patient's quality of life
  Group 1 - Participants with Conventional Twin Block appliance Group 2 - Participants with 3D printed Twin Block appliance
Masking Description: Investigator will be masked with the randomization sequance & allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Twin Block Appliance (Active Comparator): Conventional TBA fabricated with polymethylmethacrylate (PMMA)
  Interventions: Device: Conventional TBA
- 3D Printed Twin Block Appliance (Experimental): 3D Twin Block Appliance fabricated with a 3D printing resin (TR07 Graphy)
  Interventions: Device: 3D TBA

INTERVENTIONS:
Device: Conventional TBA — Conventional TBA fabricated with polymethylmethacrylate
  Arms: Conventional Twin Block Appliance
Device: 3D TBA — 3D TBA made out of a 3D printing resin (Graphy TR07)
  Arms: 3D Printed Twin Block Appliance

SUMMARY:
The Twin Block appliance is a removable orthodontic appliance that is used to help correct a backward positioned lower jaw in growing children. This appliance works by guiding the lower jaw forward to a specific position over a certain period of time. After completing the treatment, patients often experience improvements in their appearance, such as an improved bite, a more balanced facial profile and improved lip posture.

The investigators' interest is to compare two types of Twin Block appliances; traditional (conventional) and 3D-printed, by examining several factors, including the amount of bacteria that stick to them, the surface roughness, and the overall effectiveness of each type.

Surface roughness refers to the texture of the appliance's surface, which could influence how much bacteria can accumulate. Rougher surfaces may trap more bacteria, potentially leading to oral health issues such as bad breath, tooth decay, and gum problems. The study will also assess the effectiveness of both the conventional and 3D-printed Twin Block appliances, focusing on factors like how well they perform in improving jaw position and achieving the desired treatment outcomes.

Additionally, the investigators want to assess how these appliances affect the quality of life related to oral health. Participants will answer questions about their experience to help understand how the type of appliance impacts their daily lives, comfort, and overall well-being during the course of treatment.

DETAILED DESCRIPTION:
RATIONALE OF STUDY

The rationale is to explore and address concerns related to the use of 3D printed resins with the Twin Block Appliance (TBA), in comparison to the conventional materials PMMA. The surface roughness of 3D printed resins, has been reported to be different from conventional materials and has been associated with increased microbial adhesion, particularly to Candida. This raises concerns about the potential oral health risks, such as dental caries and mucosal inflammation, when using 3D printed materials for orthodontic appliances.

Based on previous literature, it is postulated that bacterial load will be present on TBA surfaces, with the possibility of variation depending on the type of material used. This study aims to determine whether the microbial load decreases or increases based on the appliance material. Till date, there still remains a research gap specifically on microbial load in Twin Block appliances, making this study relevant in understanding the risks involved in the use of different materials in orthodontics.

Additionally, the study seeks to examine the effectiveness of 3D printed TBAs in reducing overjet and improving dental aesthetics, as well as the acceptability of these appliances by patients compared to conventional TBAs.

Furthermore, the study will compare the potential complications and treatment failures between conventional and 3D printed TBAs, aiming to demonstrate the practicality and feasibility of adopting 3D printing in the digital workflow for this appliance. By focusing on microbial adherence, surface roughness, treatment effectiveness, and oral health-related quality of life (OHRQoL), the study intends to provide valuable insights that could support the adoption of 3D printing technology in orthodontics while addressing the potential oral health risks associated with its use.

PRIMARY OBJECTIVES

1. To compare the microbial adherence between the conventional Twin Block appliance (TBA) and the 3D-printed Twin Block appliance (3D TBA).
2. To compare the impact of the appliances on the perception on dental aesthetics in patients wearing the TBA and 3D TBA.

SECONDARY OBJECTIVES

1. To compare the surface roughness of TBA and 3D TBA at baseline and after 6 months.
2. To determine the association between the surface roughness of TBA and 3D TBA with microbial adherence
3. To compare the impact of the appliances on the daily performances in patients wearing the TBA and 3D TBA.
4. To compare treatment effectiveness in the time required to reduce overjet within normal limits (<4mm)
5. To compare treatment effectiveness in achieving the skeletal and dental changes between TBA and 3D TBA.
6. To compare the risks for the potential complications and treatment failures between the TBA and 3D TBA.

SAMPLE SIZE ESTIMATION Sample size was determined using G*Power Software (Version 3.1.9.2). Sample size calculation was performed based on an alpha significance level of 0.05 and an effect size of 1.316 to achieve 80% power, to detect a significant difference between the groups. Based on the calculation, the total number of participants needed for this study is 11 participants per group. To anticipate a 36% drop out rate, the sample size required would be at least 15 participants per group.

METHODOLOGY

1. Recruitment

   * Participants will be recruited from the Orthodontic Postgraduate Clinic, Faculty of Dentistry, Universiti Malaya. They must meet inclusion and exclusion criteria for the study.
   * A total of 32 participants will be enrolled, with 16 males and 16 females, ensuring that gender is accounted for in the study.
2. Block Randomization

   * Block randomization will be performed using an online block randomization list generator (www.sealedenvelope.com) by another researcher who will not be involved in the clinical procedure.
   * A list will be generated and the random allocation sequences will be kept in sealed dark envelopes, labelled for gender and numbered accordingly
   * Participants will be assigned to two groups, either conventional TBA or 3D TBA based on the random allocation sequence and will be revealed when the envelopes are opened on the day of appointment.
3. Informed consent and assent

   * Prior to participation, patients and their parents will be provided with an information sheet and will be asked to give written consent and assent in their preferred language (English or Bahasa Melayu).
   * Once consent is obtained, participants will be randomly assigned to either the TBA or 3D TBA group.

Methodology based on objectives:

Primary objective 1: To compare the microbial adherence between the conventional Twin Block appliance (TBA) and the 3D-printed Twin Block appliance (3D TBA).

* Microbial adherence will be assessed at three time points: baseline (T0), 3 months (T1), and 6 months (T2) after appliance fitting.
* At the 3rd and 6th month follow up, the upper and lower Twin Block appliances will be placed separately in plastic containers filled with brain heart infusion (BHI) broth media, using sterilized tweezers, and sonicated in a water bath to dislodge microorganisms attached to the appliances.
* After sonication, the TBA will be removed from the containers, and the dislodged microorganisms will be transported to the Microbiology Lab for further processing.
* Samples will then be vortexed and serially diluted before plating on BHI, MSA, and SDA agar plates to allow enumeration of colony-forming units (CFU).
* Incubation will take place at 37°C for 18 to 24 hours and the plates showing CFU counts between 30 to 300 will be selected for enumeration.
* The researcher will be trained and assisted by a clinical microbiologist to perform the microbial colony count.
* The analysis will be performed in a sterile environment under a Class 2 Biosafety Cabinet.

Primary Objective 2: To compare the impact of the appliances on the perception of dental aesthetics in patients wearing the TBA and 3D TBA.

* Participants will complete the Psychosocial Impact of Dental Aesthetics Questionnaire (PIDAQ) at the following time points: baseline (T0), mid-treatment (T1), post-treatment (TF), and 3 months after final treatment (TF3).
* This questionnaire will assess participants' perceptions of dental aesthetics, including their psychosocial impact, to measure the appliances' effect on their self-esteem and social interactions.
* The PIDAQ will provide an objective measure of how wearing either the conventional TBA or 3D TBA affects dental aesthetics perception.

Secondary Objective 1: To compare the surface roughness of TBA and 3D TBA at baseline and after 6 months.

* Surface roughness will be measured three times in three different directions on each appliance using a profilometer at baseline (T0) and 6 months (T2) after appliance fitting
* The three measurements performed for each specimen will be used to calculate the average surface roughness (Ra) and will be recorded in micrometres (µm).
* The surface that it captures it best recorded on a flat surface, hence, the fitting surface and biting surface on the bite blocks of the upper and lower appliance will be used as reference point as the area of interest is similar for both conventional TBA and 3D TBA.

  -- Surface roughness is crucial because rough surfaces may promote microbial adherence, influencing the results of the microbial analysis.
* These measurements will be compared between the conventional TBA and the 3D TBA to assess the impact of different materials on appliance surface texture.

Secondary Objective 2: To determine the association between the surface roughness of TBA and 3D TBA with microbial adherence.

* After measuring the surface roughness at baseline and 6 months, a correlation analysis will be performed to assess the relationship between surface roughness and microbial adherence for both TBA and 3D TBA appliances.
* This analysis will help determine whether rougher surfaces contribute to higher microbial adherence.

Secondary Objective 3: To compare the impact of the appliances on the daily performances in patients wearing the TBA and 3D TBA.

* Participants will complete the Child Oral Impacts on Daily Performances (Child-OIDP) questionnaire at baseline (T0), mid-treatment (T1), post-treatment (TF), and 3 months after final treatment (TF3).
* The Child-OIDP assesses the impact of dental appliances on daily activities such as eating, speaking, and social interactions, providing insight into the patients' quality of life during treatment.
* This will allow comparison of the effects on daily function between TBA and 3D TBA.

Secondary Objective 4: To compare treatment effectiveness in the time required to reduce overjet within normal limits (<4mm).

* The overjet and other occlusal measurements (i.e canine relationships, molar relationships and overbite) will be recorded for the participants at the start of the study (T0), and every month for six months after the initial fitting of the Twin Block appliance (T0-T6)
* The target is to reduce overjet to less than 4mm, and the appliance's efficiency in achieving this will be compared between the conventional TBA and 3D TBA.

Secondary Objective 5: To compare treatment effectiveness in achieving the skeletal and dental changes between TBA and 3D TBA.

* Once the overjet is considered clinically corrected (<4 mm) and stable, the appliance will be removed, and the treatment will be deemed complete.
* Lateral cephalometric radiographs will be taken at baseline (T0) and end of treatment (TF) to assess skeletal and dental changes.
* Measurements on the lateral cephalogram using cephalometric parameters based on Pancherz analysis will be performed using Winceph (Rise Corporation, Japan).
* This data will provide insight into the treatment outcomes and compare the efficiency of the conventional and 3D TBA.

Secondary Objective 6: To compare the risks for potential complications and treatment failures between the TBA and 3D TBA.

* The study will also record failure of treatment rates, number of routine and emergency visits, number and nature of complications.
* Participants will be considered noncompliant (treatment failure) if overjet does not reduce by at least 10% within 6 months or if overjet fails to reach normal levels (<4mm) after 12 months.
* Breakage of the appliance more than 3 times over the initial 6-month period and/ or persistent poor oral hygiene with associated harms hindering treatment progress will also be regarded as a failure
* Details of adverse events (complications) in both groups, including breakages and harms reported during routine or emergency visits, will be collected from participants' notes using a data collection sheet and categorized according to their nature and severity.

STATISTICAL ANALYSES Results obtained will be computed using Statistical Package for Social Science (SPSS) software version 29.0.1 for Mac OS Catalina. Parametric tests will be applied for normally distributed data and non-parametric tests will be applied for non-normally distributed data. The level of statistical significance will be predefined at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Class II Division 1 incisor relationship
2. Overjet of ≥ 7mm
3. Age range of children: 10-12 years in females, 12-14 years in males
4. All permanent incisors and molars erupted
5. ICDAS ≥ score 3 and BPE ≥ 3
6. Able to understand English or Bahasa Melayu

Exclusion Criteria:

1. Patients with craniofacial syndromes (example: cleft lip and palate)
2. Patients with previous history of orthodontic treatment
3. Patients with hyperdivergent facial type (MMPA > 40º)
4. Untreated gingival disease (e.g.: gingivitis, periodontitis)

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-01-17 (Estimated); Study Completion 2027-01-17 (Estimated)

PRIMARY OUTCOMES:
Microbial colony counts (CFU/ml) on the appliances. | 6 months
  Microbial colony count on the conventional Twin Block appliance & 3D printed Twin Block appliance
  The conventional Twin Block appliance (TBA) and the 3D printed Twin Block 3D TBA appliance that are collected from the patients before issue of the appliance (T0), after 3 months (T1) and at 6 months (T2). The TBA will be placed in BHI media and then will undergo the process of sonication, which will produce the bacteria suspension. This bacteria suspension will then be cultured in an agar plate with BHI media and incubated for 18 - 24 hours. The total colony per count will then be counted and recorded.
Assessment of Oral health-related quality of life (OHRQoL): PIDAQ Scores | 12 months
  The Malaysian psychosocial impact of dental aesthetics (PIDAQ) questionnaire consists of 22 questions that measures the impact of malocclusion on the dental self-confidence (DSC), social impact (SI), psychological impact (PI) and aesthetic concern (AC). The responses to each question will be scored on a 5-point Likert scale and coded as follows: 0 = Not at all; 1 = A little; 2 = Somewhat; 3 = Strongly; 4 = Very strongly. The PIDAQ questionnaire will be distributed at T0 (at baseline- at issue appointment) T1 (at 3-months) TF (Final time-point).

SECONDARY OUTCOMES:
Surface roughness (Ra) of the appliances | 6 months
  The surface roughness of both the conventional and 3D TBA appliances will be assessed using a profilometer (Mitutoyo Surf Test, Japan) at baseline and at T2 (6 months).
  Surface roughness will be assessed by measuring each specimen three times in three different directions. The three measurements performed for each specimen will be used to calculate the average surface roughness (Ra) and will be recorded in micrometres (µm).
Assessment of Oral health-related quality of life (OHRQoL): Child-ODIP (prevalence and scores) | 12 months
  The oral impacts on daily performances for children (Child-ODIP) questionnaire will evaluate oral impacts across eight performances i.e eating, speaking, cleaning teeth, relaxing, emotional stability, smiling, doing schoolwork and socialising.
  The Child-ODIP questionnaire will be distributed at T0 (at baseline- at issue appointment) T1 (at 3-months) TF3 (3-months after final time-point).
Treatment effectiveness: Treatment duration (in months) | 12 months
  The time (in months) required to reduce overjet to normal limits (<4 mm).
  The overjet and other occlusal measurements (i.e canine relationships, molar relationships and overbite) will be recorded for the participants at the start of the study (T0) , and every month after the initial fitting of the Twin Block appliance until normal overjet (2-4mm) is achieved (T0-TFinal).
Treatment effectiveness: Linear measurements (in mm) | 12 months
  A lateral cephalogram will be taken at T0 and at the end of functional appliance treatment (TFinal), which is anticipated up to 12 months, to assess for skeletal and dental changes. Measurements of sagittal changes on the lateral cephalogram will be recorded in millimeters (mm).
Frequency of the potential complications and treatment failures between the conventional Twin Block appliance and the 3D printed Twin Block appliances | 12 months
  The study will also record potential complications and treatment failures between the conventional TBA and the 3D TBA. Frequency of adverse events (complications) in both groups, including breakages and harms reported such as during routine or emergency visits, will be collected from participants' notes using a data collection sheet and categorized according to their nature and severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Orthodontic Postgraduate Clinic, Faculty of Dentistry, Universiti Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yusuf H, Gherunpong S, Sheiham A, Tsakos G. Validation of an English version of the Child-OIDP index, an oral health-related quality of life measure for children. Health Qual Life Outcomes. 2006 Jul 1;4:38. doi: 10.1186/1477-7525-4-38. PMID 16813660
- [Background] Marsh PD. Dental plaque as a biofilm and a microbial community - implications for health and disease. BMC Oral Health. 2006 Jun 15;6 Suppl 1(Suppl 1):S14. doi: 10.1186/1472-6831-6-S1-S14. PMID 16934115
- [Background] Klages U, Claus N, Wehrbein H, Zentner A. Development of a questionnaire for assessment of the psychosocial impact of dental aesthetics in young adults. Eur J Orthod. 2006 Apr;28(2):103-11. doi: 10.1093/ejo/cji083. Epub 2005 Oct 28. PMID 16257989
- [Background] Graf S, Tarraf NE, Vasudavan S. Direct printed removable appliances: A new approach for the Twin-block appliance. Am J Orthod Dentofacial Orthop. 2022 Jul;162(1):103-107. doi: 10.1016/j.ajodo.2021.08.019. PMID 35772870
- [Background] El-Huni A, Colonio Salazar FB, Sharma PK, Fleming PS. Understanding factors influencing compliance with removable functional appliances: A qualitative study. Am J Orthod Dentofacial Orthop. 2019 Feb;155(2):173-181. doi: 10.1016/j.ajodo.2018.06.011. PMID 30712688
- [Background] Mohd Tahir N, Wan Hassan WN, Saub R. Comparing retainers constructed on conventional stone models and on 3D printed models: a randomized crossover clinical study. Eur J Orthod. 2019 Aug 8;41(4):370-380. doi: 10.1093/ejo/cjy063. PMID 30321319
- [Background] Yacob N, Ahmad NA, Safii SH, Yunus N, Abdul Razak F. Is microbial adhesion affected by the build orientation of a 3-dimensionally printed denture base resin? J Prosthet Dent. 2023 Jul;130(1):131.e1-131.e7. doi: 10.1016/j.prosdent.2023.04.017. Epub 2023 May 19. PMID 37210224
- [Background] Wuersching SN, Westphal D, Stawarczyk B, Edelhoff D, Kollmuss M. Surface properties and initial bacterial biofilm growth on 3D-printed oral appliances: a comparative in vitro study. Clin Oral Investig. 2023 Jun;27(6):2667-2677. doi: 10.1007/s00784-022-04838-7. Epub 2022 Dec 28. PMID 36576565
- [Background] Belayutham S, Wan Hassan WN, Razak FA, Mohd Tahir NNZ. Microbial adherence on vacuum-formed retainers with different surface roughness as constructed from conventional stone models and 3D printed models: a randomized controlled clinical trial. Clin Oral Investig. 2023 Jun;27(6):3245-3259. doi: 10.1007/s00784-023-04940-4. Epub 2023 Mar 22. PMID 36947263
- [Background] Pacha MM, Fleming PS, Pandis N, Shagmani M, Johal A. The use of the Hanks Herbst vs Twin-block in Class II malocclusion: A randomized controlled trial. Am J Orthod Dentofacial Orthop. 2023 Sep;164(3):314-324.e1. doi: 10.1016/j.ajodo.2023.06.002. Epub 2023 Jul 4. PMID 37409988
- [Background] Farhadian N, Usefi Mashoof R, Khanizadeh S, Ghaderi E, Farhadian M, Miresmaeili A. Streptococcus mutans counts in patients wearing removable retainers with silver nanoparticles vs those wearing conventional retainers: A randomized clinical trial. Am J Orthod Dentofacial Orthop. 2016 Feb;149(2):155-60. doi: 10.1016/j.ajodo.2015.07.031. PMID 26827971